CLINICAL TRIAL: NCT05382143
Title: The Effect of Selective Oxytocin Receptor Inhibitors on Endometriosis-related Pain
Acronym: ENDOBAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL67501.091.18
Record Dates: First submitted 2022-04-13; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — atosiban

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All the participants in this pilot study will receive atosiban
  Interventions: Drug: Atosiban

INTERVENTIONS:
Drug: Atosiban — Pilot study

SUMMARY:
A pilot study to investigate the potential role of atosiban, a selective oxytocin receptor inhibitor, in the management of endometriosis-related pain. Ten patients will be administered atosiban intravenously during 6 hours on a day during their period when they experience (severe) pain

DETAILED DESCRIPTION:
Rationale: Endometriosis is a common chronic, incurable condition in which endometrium-like tissue implants outside the uterus. In the Netherlands approximately 405,000 women between 15 and 50 years of age are estimated to have endometriosis in some degree. Symptoms may vary through the menstrual cycle and include but are not limited to: dysmenorrhea (pain during menstruation), chronic pelvic pain, dyspareunia (pain during or after sexual intercourse) and dyschezia (pain during defecation). Current treatment options consist of analgesics, hormonal treatment and more or less invasive surgery. Following histological findings and in vitro and animal research, oxytocin receptor antagonists might be an alternative, non-hormonal, non-invasive treatment option. Except for one study on advanced reproductive techniques, no studies have reported the use of selective oxytocin receptor antagonists in human patients. The investigators hypothesize atosiban, a selective oxytocin receptor antagonist that is currently available in an intravenous administration form, can significantly lower patients' pain scores. If this pilot study shows atosiban is an effective treatment option for women with endometriosis, the investigators intend to develop a patient-friendly mode of administration for atosiban.

Objective: To investigate the potential of atosiban as a treatment for pain caused by endometriosis.

Study design: Phase II interventional pilot study Study population: 10 patients with laparoscopic, MRI or ultrasound proven endometriosis Intervention (if applicable): Atosiban 6,75mg intravenously bolus, followed by 18mg per hour continuous infusion for 3 hours, followed by 6mg per hour continuous infusion for 3 more hours.

Main study parameters/endpoints: Reduction in pain score (VAS), use of analgesics, experienced side effects.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will be admitted in day-care while they will receive intravenous treatment with atosiban. They will be asked to keep a menstrual diary for one month, one time before the treatment and another time afterwards. Furthermore, participants will be asked to fill in questionnaires on quality of life and their medical history. Their pain scores will be taken at several time points. The investigators will take blood samples at the start and at the end of the treatment. The most important risk for participants is the risk of side effects related to atosiban. These include nausea (>10%), headache, dizziness, flushes, tachycardia, hypotension, vomiting, hypoglycaemia and local reaction on the place of injection (1-10%). The most severe side effect described is pulmonary oedema. This was mostly in combination with other tocolytic agents and very rare, the side effects are generally considered to be mild. Atosiban has been administered on a routine basis to pregnant women with preterm labour in the same regimen as is used now. However, the investigators will administer atosiban for a shorter period of time. According to the risk classification of the Netherlands Federation of University hospitals for patients participating in this study, the risk has been assessed as "moderate".

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic, MRI or ultrasound confirmed endometriosis
* Dysmenorrhea with an average pain score ≥5 on the most painful day during menstrual period or withdrawal bleeding

Exclusion Criteria:

* Inability to come to the hospital for the experiment
* Suspicion on a (post)menopausal state
* Continuous treatment with oral contraceptives or progestagens
* Current use of gonadotrophin releasing-hormone agonist
* Current ovarian stimulation
* Current breastfeeding
* Labour or breastfeeding within the last 6 weeks
* Diagnosis of chronic pelvic pain
* Inability to give informed consent
* Language barrier
* Diabetes Mellitus, type I or II
* Hypersensitivity to atosiban or mannitol
* Use of systemic betamimetics
* Use of calcium channel blockers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in pain during and after the administration of atosiban | Change from baseline up to 4 weeks
  Pain scores on a visual analogue scale from 0 to 10, where higher scores mean more pain, during treatment and the month following treatment

SECONDARY OUTCOMES:
Side effects of atosiban | Up to 4 weeks
  Side effects may include headache, nausea and dizziness. Side effects are measured on visual analogue scale from 0 to 10, where higher scores mean more complaints.
Levels of serum prostaglandins | Baseline and directly after the administration of 6 hours atosiban
  Prostaglandin levels will be measured in blood in pg/mL
Side effect of atosiban | Baseline and directly after the administration of 6 hours atosiban
  A potential side effect of atosiban is hyperglycaemia. Glucose levels will be measured in blood in mmol/l.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No